CLINICAL TRIAL: NCT06689371
Title: Dry Needling Versus Dry Cupping on Pain and Disability in Cervicogenic Headache Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Samara Elsaeed Shahen, Demonstrater, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.T.REC/012/005277
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Dry Needling; Dry Cupping; Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Dry needling): The 15 patients will receive three dry needling sessions per week for four (Experimental)
  Interventions: Other: Group A (Dry Needling)
- Group B (Dry cupping): The 15 patients will receive three dry cupping sessions per week for four we (Experimental)
  Interventions: Other: Group B (Dry cupping)
- Group C (control): The 15 patients will receive standard exercise three sessions per week for four w (Active Comparator)
  Interventions: Other: Group C (control)

INTERVENTIONS:
Other: Group A (Dry Needling) — The patient will receive dry needling on suboccipital, upper trapezius and SCM muscles with conventional therapy 3 sessions per week for 4 weeks.
  Arms: Group A (Dry needling): The 15 patients will receive three dry needling sessions per week for four
Other: Group B (Dry cupping) — Patients will receive dry cupping on suboccipital, upper trapezius and SCM muscles weeks with conventional therapy 3 sessions per week for 4 weeks.
  Arms: Group B (Dry cupping): The 15 patients will receive three dry cupping sessions per week for four we
Other: Group C (control) — will receive standard exercise three sessions per week for four weeks. This standard regimen consists of the same exercises as group A and B.
  Arms: Group C (control): The 15 patients will receive standard exercise three sessions per week for four w

SUMMARY:
This study aims to compare the added effects of dry needling and dry cupping to conventional physical therapy on headache pain intensity, headache frequency, headache duration, upper cervical range of motion, and disability levels in patients with cervicogenic headache.

It will be assumed that:

* All patients will follow all the given instructions strictly during the study duration, regarding the assessment and the treatment procedure.
* All participants will be evaluated under the same environmental conditions.

DETAILED DESCRIPTION:
Neck pain is a highly popular musculoskeletal complain and the second most common musculoskeletal condition affecting people in their adolescence after low back pain. It is a common condition affecting general populations with high economic burden for neck pain including raised treatment costs, reduced productivity, and job-related problems. Headache is one of the most common disorders associated with neck pain with a potential for major disability.

Migraine, tension-type headache (TTH), and cervicogenic headache (CGH) are common types of headaches that negatively affect the quality of life, work activities, and family life. It has a direct or indirect economic burden on society.

Cervicogenic headache (CH) is a secondary headache caused by a disorder of the cervical spine and its disc or bony and/or periarticular components. In this type, pain originates from the back of neck and radiates towards the front of the head and eye on the same side. CGH can last from a few hours to days. The prevalence rate of CGH was estimated to be from 0.4% to 2.5% in the adult population and appears to affect women more than men.

The physiological mechanism of pain in CGH headache is the convergence of upper cervical spinal nerves (C1, C2, and C3) afferents and trigeminal afferents in the trigeminocervical nucleus caudalis. This convergence allows the bidirectional referral of painful sensations between the neck and trigeminal sensory receptive fields of the face and head.

Another cause of CGH is myofascial trigger points in the muscles. These trigger points, which are innervated by C1 to C3 (specifically in the suboccipital, semispinalis capitis, splenius cervices, trapezius, and sternocleidomastoid), can cause referral pain in various parts of the head.

Systematic review concluded that patients with CGH have significantly decreased cervical ROM and muscle function. Those patients have deep neck flexor weakness and tightness of the Sternocleidomastoid (SCM), trapezius and other muscles in the scapular region.

Management of CGH can involve a wide variety of therapeutic techniques, including medication, anesthetic and corticosteroid blocks, pulsed radiofrequency, cognitive therapy, relaxation therapy and physical therapy. Physical therapy interventions are recommended as nonpharmacological approaches for the treatment of CGH patients. These interventions include spinal manipulation, mobilization, manual therapy, dry needling, and therapeutic exercise.

Dry needling (DN) is an intervention method commonly used by physiotherapists for treatment of muscle pain associated with Trigger points (TrPsA). Acupuncture needles are placed directly into Muscle Trigger points (MTrPs) during this minimally invasive treatment. The benefits of DN include immediate relief in local, referred, and widespread pain and a restoration of range of motion and muscle activation patterns.

A previous study reported that the DN into the MTrPs of the suboccipital and upper trapezius muscles decreased headache index (HI), MTrP tenderness, increased functional rating index, and the range of motions in patients with CGH.

Cupping therapy (CT) is a physical traditional Chinese medicine (TCM) practiced by ancient Chinese, Egyptians, and Greeks and currently used by therapists and acupuncturists in the treatment of a wide range of medical conditions and played a vital role in human health. This alternative therapy involves creating a vacuum inside a cup positioned over the surface of the skin, using the local negative pressure to improve blood flow.

It has been used to treat various medical conditions, such as musculoskeletal injuries, dermatologic conditions, and chemical imbalances within the body. The most common use is reducing musculoskeletal or myofascial pain. It has been used to treat fibromyalgia, rheumatoid arthritis, neck and shoulder pain, and low back pain.

Cupping produces localized hyperemia to the applied area, The dilation of capillaries improves microcirculation which decreases muscle tone and promotes healing via metabolic changes.

Cupping therapy was the most preferred treatment method after herbal treatments in headache patients. Acupuncture and wet cupping method has a beneficial effect on pain intensity and cervical ROM in cervical headache patients when compared to shame acupuncture.

Moreover, a systematic review concluded that the evidence for dry needling and cupping is not greater than placebo in treatment of myofascial pain.

There is no study compare between effect of dry needling and dry cupping on cervicogenic headache patients.

Therefore, this study aims to compare between the effect of dry needling versus dry cupping on pain, Range of Motion (ROM) and level of disabilities in patients of cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be included in our study if they meet the following criteria:

  * Age between 25-45 years old for both genders.
  * No physiotherapy intervention for the last three months.
  * Intermittent headaches of varying duration and pain level at the rate of one headache per week for greater than 2 months.
  * Ipsilateral neck, shoulder, or arm pain.
  * Provocation of usual head pain by neck movement, sustained awkward neck positions or external pressure over the upper cervical or occipital region on the symptomatic side.
  * Limited neck ROM > 10 degrees confirmed by a positive Flexion Rotation Test.
  * Active trigger points (TrPs) within the suboccipital, upper trapezius or sternocleidomastoid muscles.

The diagnosis of active TrPs will be based on the major criteria proposed by):

* Presence of a palpable taut band in a skeletal muscle
* presence of a hypersensitive point in the taut band
* local twitch response elicited by the snapping palpation of the taut band
* reproduction of the referred pain in response to compression
* patient recognition of the referred pain as a familiar symptom

Exclusion Criteria:

* The patients will be excluded if they have:

  * Cervical radiculopathy.
  * History of neck, shoulder trauma or surgery.
  * Physical therapy intervention in the neck and shoulder region in the previous 3 months.
  * Vertebrobasilar insufficiency or vestibular dysfunctions.
  * Evidence of cognitive deficits.
  * Presence of any needle contraindication.
  * Presence of any cupping contraindication.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-13 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion (CROM) | Pre- intervention and after 4 weeks of treatment
  CROM device will be used for the assessment of upper cervical ROM.
The Arabic Version Of Neck Disability Index (NDI). | Pre- intervention and after 4 weeks of treatment
  to assess the level of disabilities in patients with cervicogenic headache, in % points.
Headache impact test 6 items | Pre- intervention and after 4 weeks of treatment
  used to assess headache severity.
Numerical pain rating scale | Pre- intervention and after 4 weeks of treatment
  used to assess headache pain intenisty.
Pressure Algometer | Pre- intervention and after 4 weeks of treatment
  used to assess trigger points pain pressure threshold

REFERENCES:
- [Background] Ahmed SM, Madbouly NH, Maklad SS, Abu-Shady EA. Immunomodulatory effects of blood letting cupping therapy in patients with rheumatoid arthritis. Egypt J Immunol. 2005;12(2):39-51. PMID 17977209
- [Background] Al-Bedah AMN, Elsubai IS, Qureshi NA, Aboushanab TS, Ali GIM, El-Olemy AT, Khalil AAH, Khalil MKM, Alqaed MS. The medical perspective of cupping therapy: Effects and mechanisms of action. J Tradit Complement Med. 2018 Apr 30;9(2):90-97. doi: 10.1016/j.jtcme.2018.03.003. eCollection 2019 Apr. PMID 30963043
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Berger AA, Liu Y, Mosel L, Champagne KA, Ruoff MT, Cornett EM, Kaye AD, Imani F, Shakeri A, Varrassi G, Viswanath O, Urits I. Efficacy of Dry Needling and Acupuncture in the Treatment of Neck Pain. Anesth Pain Med. 2021 Apr 3;11(2):e113627. doi: 10.5812/aapm.113627. eCollection 2021 Apr. PMID 34336626
- [Background] Bravo Petersen SM, Vardaxis VG. The flexion-rotation test performed actively and passively: a comparison of range of motion in patients with cervicogenic headache. J Man Manip Ther. 2015 May;23(2):61-7. doi: 10.1179/2042618614Y.0000000085. PMID 26109826
- [Background] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Background] Cardoso R, Seixas A, Rodrigues S, Moreira-Silva I, Ventura N, Azevedo J, Monsignori F. The effectiveness of Sustained Natural Apophyseal Glide on Flexion Rotation Test, pain intensity, and functionality in subjects with Cervicogenic Headache: A Systematic Review of Randomized Trials. Arch Physiother. 2022 Sep 1;12(1):20. doi: 10.1186/s40945-022-00144-3. PMID 36045409
- [Background] Chys M, De Meulemeester K, De Greef I, Murillo C, Kindt W, Kouzouz Y, Lescroart B, Cagnie B. Clinical Effectiveness of Dry Needling in Patients with Musculoskeletal Pain-An Umbrella Review. J Clin Med. 2023 Feb 2;12(3):1205. doi: 10.3390/jcm12031205. PMID 36769852
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Ekhator C, Urbi A, Nduma BN, Ambe S, Fonkem E. Safety and Efficacy of Radiofrequency Ablation and Epidural Steroid Injection for Management of Cervicogenic Headaches and Neck Pain: Meta-Analysis and Literature Review. Cureus. 2023 Feb 13;15(2):e34932. doi: 10.7759/cureus.34932. eCollection 2023 Feb. PMID 36938280
- [Background] Fernandez-de-las-Penas C, Cuadrado ML, Arendt-Nielsen L, Simons DG, Pareja JA. Myofascial trigger points and sensitization: an updated pain model for tension-type headache. Cephalalgia. 2007 May;27(5):383-93. doi: 10.1111/j.1468-2982.2007.01295.x. Epub 2007 Mar 14. PMID 17359516
- [Background] France S, Bown J, Nowosilskyj M, Mott M, Rand S, Walters J. Evidence for the use of dry needling and physiotherapy in the management of cervicogenic or tension-type headache: a systematic review. Cephalalgia. 2014 Oct;34(12):994-1003. doi: 10.1177/0333102414523847. Epub 2014 Mar 12. PMID 24623124
- [Background] Ge W, Leson C, Vukovic C. Dry cupping for plantar fasciitis: a randomized controlled trial. J Phys Ther Sci. 2017 May;29(5):859-862. doi: 10.1589/jpts.29.859. Epub 2017 May 16. PMID 28603360
- [Background] Ghods R, Sayfouri N, Ayati MH. Anatomical Features of the Interscapular Area Where Wet Cupping Therapy Is Done and Its Possible Relation to Acupuncture Meridians. J Acupunct Meridian Stud. 2016 Dec;9(6):290-296. doi: 10.1016/j.jams.2016.06.004. Epub 2016 Sep 15. PMID 28010830
- [Background] Gugliotti M, Tau J, Gallo K, Sagliocca N, Horan M, Sussman N, Wisnewski R. Between-week reliability of the cervical range of motion (CROM) device for upper cervical rotation. J Man Manip Ther. 2021 Jun;29(3):176-180. doi: 10.1080/10669817.2020.1805691. Epub 2020 Aug 18. PMID 32808588
- [Background] Iglesias-Gonzalez JJ, Munoz-Garcia MT, Rodrigues-de-Souza DP, Alburquerque-Sendin F, Fernandez-de-Las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in patients with chronic nonspecific low back pain. Pain Med. 2013 Dec;14(12):1964-70. doi: 10.1111/pme.12224. Epub 2013 Aug 15. PMID 23947760
- [Background] Ireland J, Window P, O'Leary SP. The impact of exercise intended for fitness or sport on the prevalence of non-specific neck pain in adults: A systematic review. Musculoskeletal Care. 2022 Jun;20(2):229-244. doi: 10.1002/msc.1592. Epub 2021 Sep 29. PMID 34586706
- [Background] Jung A, Carvalho GF, Szikszay TM, Pawlowsky V, Gabler T, Luedtke K. Physical Therapist Interventions to Reduce Headache Intensity, Frequency, and Duration in Patients With Cervicogenic Headache: A Systematic Review and Network Meta-Analysis. Phys Ther. 2024 Feb 1;104(2):pzad154. doi: 10.1093/ptj/pzad154. PMID 37941472
- [Background] Kietrys DM, Palombaro KM, Azzaretto E, Hubler R, Schaller B, Schlussel JM, Tucker M. Effectiveness of dry needling for upper-quarter myofascial pain: a systematic review and meta-analysis. J Orthop Sports Phys Ther. 2013 Sep;43(9):620-34. doi: 10.2519/jospt.2013.4668. PMID 23756457
- [Background] Kim JI, Lee MS, Lee DH, Boddy K, Ernst E. Cupping for treating pain: a systematic review. Evid Based Complement Alternat Med. 2011;2011:467014. doi: 10.1093/ecam/nep035. Epub 2011 Jun 23. PMID 19423657
- [Background] Misailidou V, Malliou P, Beneka A, Karagiannidis A, Godolias G. Assessment of patients with neck pain: a review of definitions, selection criteria, and measurement tools. J Chiropr Med. 2010 Jun;9(2):49-59. doi: 10.1016/j.jcm.2010.03.002. PMID 21629550
- [Background] Mohamed AA, Shendy WS, Semary M, Mourad HS, Battecha KH, Soliman ES, Sayed SHE, Mohamed GI. Combined use of cervical headache snag and cervical snag half rotation techniques in the treatment of cervicogenic headache. J Phys Ther Sci. 2019 Apr;31(4):376-381. doi: 10.1589/jpts.31.376. Epub 2019 Apr 1. PMID 31037013
- [Background] Mousavi-Khatir SR, Fernandez-de-Las-Penas C, Saadat P, Javanshir K, Zohrevand A. The Effect of Adding Dry Needling to Physical Therapy in the Treatment of Cervicogenic Headache: A Randomized Controlled Trial. Pain Med. 2022 Mar 2;23(3):579-589. doi: 10.1093/pm/pnab312. PMID 34687308
- [Background] Murtza S, Noor R, Bashir MS, Ikram M. Effects of sustained natural apophyseal glides versus rocabado 6 x 6 program in subjects with cervicogenic headache. BMC Musculoskelet Disord. 2024 Feb 22;25(1):169. doi: 10.1186/s12891-024-07290-8. PMID 38389050
- [Background] Nunez-Cabaleiro P, Leiros-Rodriguez R. Effectiveness of manual therapy in the treatment of cervicogenic headache: A systematic review. Headache. 2022 Mar;62(3):271-283. doi: 10.1111/head.14278. Epub 2022 Mar 16. PMID 35294051
- [Background] Ogince M, Hall T, Robinson K, Blackmore AM. The diagnostic validity of the cervical flexion-rotation test in C1/2-related cervicogenic headache. Man Ther. 2007 Aug;12(3):256-62. doi: 10.1016/j.math.2006.06.016. Epub 2006 Nov 16. PMID 17112768
- [Background] Polat B, Saatci O, Yilmaz NH, Duz OA. The frequency of complementary and integrative medicine methods in headache patients and their spending habits. Neurol Neurochir Pol. 2018 May-Jun;52(3):347-351. doi: 10.1016/j.pjnns.2017.12.007. Epub 2017 Dec 24. PMID 29306601
- [Background] Pourahmadi M, Dommerholt J, Fernandez-de-Las-Penas C, Koes BW, Mohseni-Bandpei MA, Mansournia MA, Delavari S, Keshtkar A, Bahramian M. Dry Needling for the Treatment of Tension-Type, Cervicogenic, or Migraine Headaches: A Systematic Review and Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab068. doi: 10.1093/ptj/pzab068. PMID 33609358
- [Background] Racicki S, Gerwin S, Diclaudio S, Reinmann S, Donaldson M. Conservative physical therapy management for the treatment of cervicogenic headache: a systematic review. J Man Manip Ther. 2013 May;21(2):113-24. doi: 10.1179/2042618612Y.0000000025. PMID 24421621
- [Background] Rendas-Baum R, Yang M, Varon SF, Bloudek LM, DeGryse RE, Kosinski M. Validation of the Headache Impact Test (HIT-6) in patients with chronic migraine. Health Qual Life Outcomes. 2014 Aug 1;12:117. doi: 10.1186/s12955-014-0117-0. PMID 25080874
- [Background] Satpute K, Nalband S, Hall T. The C0-C2 axial rotation test: normal values, intra- and inter-rater reliability and correlation with the flexion rotation test in normal subjects. J Man Manip Ther. 2019 May;27(2):92-98. doi: 10.1080/10669817.2018.1533195. Epub 2018 Oct 12. PMID 30935342
- [Background] Sedighi A, Nakhostin Ansari N, Naghdi S. Comparison of acute effects of superficial and deep dry needling into trigger points of suboccipital and upper trapezius muscles in patients with cervicogenic headache. J Bodyw Mov Ther. 2017 Oct;21(4):810-814. doi: 10.1016/j.jbmt.2017.01.002. Epub 2017 Jan 6. PMID 29037632
- [Background] Shen WC, Jan YK, Liau BY, Lin Q, Wang S, Tai CC, Lung CW. Effectiveness of self-management of dry and wet cupping therapy for low back pain: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Dec 23;101(51):e32325. doi: 10.1097/MD.0000000000032325. PMID 36595746
- [Background] Shimohata K, Hasegawa K, Onodera O, Nishizawa M, Shimohata T. The Clinical Features, Risk Factors, and Surgical Treatment of Cervicogenic Headache in Patients With Cervical Spine Disorders Requiring Surgery. Headache. 2017 Jul;57(7):1109-1117. doi: 10.1111/head.13123. Epub 2017 Jun 5. PMID 28581034
- [Background] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- [Background] Stephens SL, Selkow NM, Hoffman NL. Dry Cupping Therapy for Improving Nonspecific Neck Pain and Subcutaneous Hemodynamics. J Athl Train. 2020 Jul 1;55(7):682-690. doi: 10.4085/1062-6050-236-19. PMID 32556324
- [Background] Mohammadi Z, Shafizadegan Z, Tarrahi MJ, Taheri N. The Effectiveness of Sternocleidomastoid Muscle Dry Needling in Patients with Cervicogenic Headache. Adv Biomed Res. 2021 Feb 26;10:10. doi: 10.4103/abr.abr_138_20. eCollection 2021. PMID 33959567
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Wood S, Fryer G, Tan LLF, Cleary C. Dry cupping for musculoskeletal pain and range of motion: A systematic review and meta-analysis. J Bodyw Mov Ther. 2020 Oct;24(4):503-518. doi: 10.1016/j.jbmt.2020.06.024. Epub 2020 Jul 30. PMID 33218554
- [Background] Yanase K, Ikezoe T, Nakamura M, Saeki J, Yagi M, Hirono T, Tamezawa T, Motomura Y, Ibuki S, Ichihashi N. Effective muscle elongation positions for the neck extensor muscles: An ultrasonic shear wave elastography study. J Electromyogr Kinesiol. 2021 Oct;60:102569. doi: 10.1016/j.jelekin.2021.102569. Epub 2021 Jun 17. PMID 34298283
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Background] Yehoshua I, Rimon O, Mizrahi Reuveni M, Peleg R, Adler L. Dry needling for the treatment of acute myofascial pain syndrome in general practitioners' clinics: a cohort study. BMC Prim Care. 2022 Dec 27;23(1):339. doi: 10.1186/s12875-022-01951-0. PMID 36572860
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800